CLINICAL TRIAL: NCT00811707
Title: To Compare Epidural Sonoanatomy Between Parturient and Non-Pregnant Young Female in Chinese Population
Brief Title: Epidural Sonoanatomy Between Parturient and Non-Pregnant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Koung-Shing Chu, Departmrnt of anesthesiology, Kaohsiung Medical University Chung-Ho Hospital
Other Study IDs: KMUH-IRB-970112
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-08

CONDITIONS: Parturients
Keywords: ultrasound image; epidural space

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: volunteers: non-pregnant female
- 2: parturients: parturients was scheduled to receive lumbar epidurals for elective cesaeran delivery labor analgesia

SUMMARY:
The failure in indwelling epidural catheter for a parturient might cause an anesthetic difficulty. Furthermore, no one can predict the accuracy of needle placement prior to skin puncture with any of landmark-based technique. This may result in multiple trying attempts at needle puncture, pain and discomforts of patients and poor patient satisfaction. The aim of this study was to explore the difference of epidural space between parturient and non-pregnant women by assessing ultrasound image.

DETAILED DESCRIPTION:
We will enroll 30 non-pregnant female volunteers and 30 parturients(ASA I-III) underwent epidural blocks. A low frequency ultrasound (2-5 MHz) with a curved array transducer is used to obtain spinal sonography for each subject. The paramedian axis was used to obtain optimal ultrasound image for spinal sonography. Outcome was evaluated by the diameter and depth of epidural space at three lumbar interspaces. Paired T-test was carried out to evaluate the statistical significance of epidual diameter and depth.

ELIGIBILITY:
Inclusion Criteria:

* parturients scheduled to receive lumbar epidurals for elective cesaeran delivery labor analgesia

Exclusion Criteria:

* Pregancy induced hypertension gestational Diabetes patients who refuse

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: from Kaohsiung Medical University Hospiral ward parturients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Hospital, Kaohsiung City, Taiwan